CLINICAL TRIAL: NCT01632306
Title: Phase I/II Study of LY2090314 and Chemotherapy in Metastatic Pancreatic Cancer Patients With Metastases Amenable to Biopsy
Brief Title: A Study of LY2090314 and Chemotherapy in Participants With Metastatic Pancreatic Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study has been terminated due to slow enrollment.
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14453; I2H-MC-JWYD (Other: Eli Lilly and Company); NCT01671202 (obsolete NCT alias)
Record Dates: First submitted 2012-06-28; First posted 2012-07-02 (Estimated); Results first posted 2018-11-19 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — 3-(9-fluoro-2-(piperidin-1-ylcarbonyl)-1,2,3,4-tetrahydro(1,4)diazepino(6,7,1-hi)indol-7-yl)-4-imidazo(1,2-a)pyridin-3-yl-1H-pyrrole-2,5-dione; Folfox protocol; Leucovorin; Fluorouracil; Oxaliplatin; Gemcitabine; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- LY2090314 + Gemcitabine (Experimental): LY2090314 given intravenously (IV) on days 1 (at cycle 1 LY2090314 given on day 0 instead of day 1), 8 and 15 in 28 day cycle in combination with 1000 milligram/square meter (mg/m^2) gemcitabine given IV on days 1, 8 and 15. Cohort closed to new enrollment per protocol addendum.
  Interventions: Drug: LY2090314; Drug: Gemcitabine
- LY2090314 + FOLFOX (Experimental): LY2090314 given IV on days 1 (at cycle 1 LY2090314 given on day 0 instead of day 1), and 15 in 28 day cycle in combination with FOLFOX (leucovorin + 5-fluorouracil + oxaliplatin) given IV, on days 1 and 15 in 28 day cycle.
  Interventions: Drug: LY2090314; Drug: FOLFOX
- LY2090314 + Gemcitabine + Nab-paclitaxel (Experimental): LY2090314 given IV on days 1 (at cycle 1 LY2090314 given on day 0 instead of day 1), 8 and 15 in 28 day cycle in combination with 1000 mg/m^2 gemcitabine + 125 mg/m^2 nab-paclitaxel given IV on days 1, 8 and 15 in 28-day cycle. New cohort opened per protocol amendment.
  Interventions: Drug: LY2090314; Drug: Gemcitabine; Drug: Nab-paclitaxel

INTERVENTIONS:
Drug: LY2090314 — LY2090314 administered IV
Drug: FOLFOX — FOLFOX administered IV
  Other Names: FOLFOX (leucovorin + 5-fluorouracil + oxaliplatin)
  Arms: LY2090314 + FOLFOX
Drug: Gemcitabine — Gemcitabine administered IV
  Other Names: Gemzar; LY188011
  Arms: LY2090314 + Gemcitabine; LY2090314 + Gemcitabine + Nab-paclitaxel
Drug: Nab-paclitaxel — Nab-paclitaxel administered IV
  Arms: LY2090314 + Gemcitabine + Nab-paclitaxel

SUMMARY:
Purpose of this phase I/II study is to test how well LY2090314 works in combination with different chemotherapies in treating participants with metastatic pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic pancreatic cancer with metastases amenable to biopsy
* Willingness to provide tissue and blood samples for research purposes
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0 or 1

Exclusion Criteria:

* History of islet cell, acinar cell, or cystadenocarcinomas
* Prior cytotoxic chemotherapy for metastatic disease, except prior gemcitabine or FOLFIRINOX (5FU + leucovorin + irinotecan + oxaliplatin)
* Radiation therapy, immunotherapy or biologic therapy <28 days prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- United States (2):
  - Mayo Clinic of Jacksonville, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota

RESULTS

PARTICIPANT FLOW:
Groups:
- LY2090314 + Gemcitabine: LY2090314 given intravenously (IV) on days 1 (at cycle 1 LY2090314 given on day 0 instead of day 1), 8 and 15 in 28 day cycle in combination with 1000 milligram/square meter (mg/m²) gemcitabine given IV on days 1, 8 and 15. Cohort closed to new enrollment per protocol addendum.
- LY2090314 + Gemcitabine + Nab-paclitaxel: LY2090314 given IV on days 1 (at cycle 1 LY2090314 given on day 0 instead of day 1), 8 and 15 in 28 day cycle in combination with 1000 mg/m² gemcitabine + 125 mg/m² nab-paclitaxel given IV on days 1, 8 and 15 in 28-day cycle. New cohort opened per protocol amendment.
Period: Overall Study
Arm/Group | LY2090314 + Gemcitabine | LY2090314 + FOLFOX | LY2090314 + Gemcitabine + Nab-paclitaxel
Started | 3 | 10 | 0
Received at Least One Dose of Study Drug | 3 | 10 | 0
Completed | 2 | 10 | 0
Not Completed | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | LY2090314 + Gemcitabine | LY2090314 + FOLFOX | Total
Number analyzed (Participants) | 3 | 10 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.7 (8.5) | 64.0 (4.9) | 63.2 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5
  Male | 2 | 6 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 8 | 11
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 9 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 3 | 10 | 13

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 4 Hours Post-Treatment on Day 0 in Glycogen Synthase Phosphorylation
Description: Change in the phosphorylation level of glycogen synthase, a glycogen synthase kinase-3 beta (GSK-3beta) inhibitor, from baseline to 4 hours post-treatment on day 0 using tumor tissue and blood specimens.
Time Frame: Baseline, 4 Hours Post-Treatment on Day 0
Population: Zero participants analyzed. GSK3β phosphorylation levels were not determined, and the primary endpoint was not examined as there wasn't viable tumor tissue for analysis.
Arm/Group | LY2090314 + Gemcitabine | LY2090314 + FOLFOX
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Overall Survival (OS)
Time Frame: Baseline to Date of Death Due to any Cause Up to 21 Months
Population: All the participants that received at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | LY2090314 + Gemcitabine | LY2090314 + FOLFOX
Number analyzed (Participants) | 3 | 10
Months | 1.8 [1.3 to 1.9] | 7.7 [2.9 to 21.2]

3. Secondary Outcome: Percentage of Participants Who Survived at 6 Months
Time Frame: Baseline to Date of Death to any cause Up to 6 Months
Population: All participants who received at least one dose of study drug.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | LY2090314 + Gemcitabine | LY2090314 + FOLFOX
Number analyzed (Participants) | 3 | 10
Percentage of participants | 0 [0 to 0] | 50.0 [26.9 to 92.9]

4. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was as the time from enrollment to the earliest documented evidence of disease progression or death,whatever comes first.
Time Frame: Baseline to Disease Progression Up to 18 Months
Population: All participants who received at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | LY2090314 + Gemcitabine | LY2090314 + FOLFOX
Number analyzed (Participants) | 3 | 10
Months | 1.8 [1.3 to 1.9] | 3.4 [2.3 to 17.5]

5. Secondary Outcome: Percentage of Participants With Complete Response (CR) or Partial Response (PR) [Overall Response Rate (ORR)]
Description: Response was defined using Response Evaluation Criteria In Solid Tumors (RECIST v1.1) criteria. CR was defined as the disappearance of all target and non-target lesions and all target and non-target lymph nodes were non-pathological or normal in size [<10 millimeter (mm) short axis]. PR was defined as having at least a 30% decrease in sum of longest diameter of target lesions taking as reference the baseline sum diameters. ORR calculated as: (sum of the number of participants with PRs and CRs) divided by (number of evaluable participants) multiplied by 100.
  A CR or PR noted as the objective status on 2 consecutive evaluations at least 4 weeks apart.
Time Frame: Baseline Up to 6 Months
Population: All participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | LY2090314 + Gemcitabine | LY2090314 + FOLFOX
Number analyzed (Participants) | 3 | 10
Percentage of Participants | 0 [NA to NA] — There were "0" participants with CR or PR. | 10.0 [0.3 to 44.5]

ADVERSE EVENTS:
Description: All participants who received at least one dose of study drug.
Arm/Group | LY2090314 + Gemcitabine | LY2090314 + FOLFOX
Serious Adverse Events (participants affected / at risk) | 3/3 | 7/10
Other Adverse Events (participants affected / at risk) | 2/3 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2090314 + Gemcitabine (N=3) | LY2090314 + FOLFOX (N=10)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gallbladder obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1)
Gastric fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Failure to Thrive (General disorders) | 0 (0) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Clostridium difficle infection (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 2 (3)
Peritoneal infection (Infections and infestations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (3)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2090314 + Gemcitabine (N=3) | LY2090314 + FOLFOX (N=10)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 8 (25)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1)
Akathisia (Nervous system disorders) | 0 (0) | 1 (7)
Alanine aminotransferase (Investigations) | 1 (1) | 4 (11)
Alkaline phosphatase (Investigations) | 0 (0) | 3 (7)
Allergic reaction (Immune system disorders) | 0 (0) | 1 (2)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (6)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (6)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 2 (3)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 4 (14)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Ascites (Gastrointestinal disorders) | 0 (0) | 2 (4)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 4 (8)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 0 (0) | 1 (6)
Cardiac troponin T increased (Investigations) | 0 (0) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 3 (13)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (5)
Creatinine increased (Investigations) | 0 (0) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 4 (14)
Dizziness (Nervous system disorders) | 0 (0) | 1 (7)
Dysgeusia (Nervous system disorders) | 0 (0) | 2 (10)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (9)
ECG QT corrected interval prolonged (Investigations) | 1 (1) | 5 (5)
Edema limbs (General disorders) | 0 (0) | 1 (2)
Edema trunk (General disorders) | 0 (0) | 1 (1)
Esophageal pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 0 (0) | 9 (30)
Fever (General disorders) | 1 (1) | 1 (4)
Flatulence (Gastrointestinal disorders) | 0 (0) | 2 (8)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (9)
night sweats (General disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (7)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 2 (8)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 2 (5)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 2 (8)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Elevated lactic acid (Investigations) | 0 (0) | 1 (1)
Mucosal infection (Infections and infestations) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 3 (9)
Nausea (Gastrointestinal disorders) | 2 (2) | 6 (26)
Death due to disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 3 (10)
Pain (General disorders) | 0 (0) | 2 (3)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (7)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 4 (21)
Platelet count decreased (Investigations) | 0 (0) | 5 (23)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (8)
White blood cell (Investigations) | 0 (0) | 1 (6)

LIMITATIONS AND CAVEATS:
Study was terminated due to slow enrollment. No participants were enrolled in arm LY2090314 + Gemcitabine + Nab-paclitaxel due to inability to enroll participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days